CLINICAL TRIAL: NCT03683433
Title: Phase II Study of the Targeted Mutant IDH2 Inhibitor Enasidenib in Combination With Azacitidine for Relapsed/Refractory AML
Brief Title: Enasidenib and Azacitidine in Treating Patients With Recurrent or Refractory Acute Myeloid Leukemia and IDH2 Gene Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0499; NCI-2018-01919 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0499 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Bilineal Leukemia; Acute Biphenotypic Leukemia; Chronic Myelomonocytic Leukemia; IDH2 Gene Mutation; Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; 2-Propanol; methanesulfonic acid; enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacitidine, enasidenib mesylate) (Experimental): Patients receive azacitidine SC or IV over 30 minutes on days 1-7 and enasidenib mesylate PO QD beginning on day 1. Cycles repeat every 4-6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Enasidenib Mesylate

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Enasidenib Mesylate — Given PO
  Other Names: 2-Methyl-1-[(4-[6-(trifluoromethyl)pyridin-2-yl]-6-{[2-(trifluoromethyl)pyridin-4-yl]amino}-1,3,5-triazin-2-yl)amino]propan-2-ol Methanesulfonate; 2-Propanol, 2-Methyl-1-((4-(6-(trifluoromethyl)-2-pyridinyl)-6-((2-(trifluoromethyl)-4-pyridinyl)amino)-1,3,5-triazin-2-yl)amino)-, Methanesulfonate (1:1); AG-221 Mesylate; CC-90007; Enasidenib Methanesulfonate; Idhifa

SUMMARY:
This phase II trial studies how well enasidenib and azacitidine work in treating patients with IDH2 gene mutation and acute myeloid leukemia that has come back (recurrent) or does not respond to treatment (refractory). Enasidenib and azacitidine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical activity of enasidenib mesylate (AG221, IDHIFA) in combination with azacitidine (AZA) for patients with relapsed/refractory acute myeloid leukemia is measured by overall response rate (ORR).

SECONDARY OBJECTIVES:

I. To determine duration of response, event-free survival (EFS), and overall survival (OS).

II. To determine the safety of enasidenib in combination with azacitidine in patients with relapsed/refractory acute myeloid leukemia (AML).

EXPLORATORY OBJECTIVES:

I. To evaluate occurrence of minimal residual disease (MRD) negative status by IDH2 mutation analysis and flow cytometry.

II. To investigate possible relationships between baseline protein and gene expression signatures and mutation profile and clinical response to the combination.

III. To evaluate the incidence and characteristics of IDH-inhibitor related differentiation syndrome (IDH-DS) with combination therapy.

OUTLINE:

Patients receive azacitidine subcutaneously (SC) or intravenously (IV) over 30 minutes on days 1-7 and enasidenib mesylate orally (PO) once daily (QD) beginning on day 1. Cycles repeat every 4-6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML or biphenotypic or bilineage leukemia (including a myeloid component) who have failed prior therapy. Patients with isolated extramedullary AML are eligible. The World Health Organization (WHO) classification will be used for AML
* Elderly (> 60 years old) patients with newly diagnosed AML not eligible for intensive chemotherapy are also eligible
* AML patients with prior history of myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) regardless of prior therapy received, are eligible at the time of diagnosis of AML
* Subjects must have documented IDH2 gene mutation
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Adequate renal function including creatinine < 2 unless related to the disease
* Total bilirubin < 2 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) < 3 x ULN unless considered due to leukemic involvement
* Provision of written informed consent
* Oral hydroxyurea and/or cytarabine (up to 2 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the principal investigator (PI). Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment

Exclusion Criteria:

* Patients with t(15;17) karyotypic abnormality or acute promyelocytic leukemia (French-American-British [FAB] class M3-AML)
* Active and uncontrolled comorbidities including active uncontrolled infection, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association (NYHA) class III/IV, clinically significant and uncontrolled arrhythmia as judged by the treating physician
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-18 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 5 years
  The study will estimate the ORR for the combination treatment, along with the Bayesian 95% credible interval. ORR will be defined as the proportion of patients who had CR (complete remission), CRh (complete remission with incomplete hematologic recovery), CRi (complete remission with incomplete count recovery), PR (partial response), and/or marrow clearance of blasts (MLFS).

SECONDARY OUTCOMES:
Event-free survival | Up to 5 years
  Kaplan-Meier method will be used to estimate the probabilities of event-free survival.
Overall survival (OS) | Up to 5 years
  Kaplan-Meier method will be used to estimate the probabilities of overall survival.
Disease-free survival (DFS) | Up to 5 years
  Log-rank tests will be used to compare among subgroups of patients in terms of DFS or OS.
Duration of response | Up to 5 years
  Log-rank tests will be used.
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 5 years

OTHER OUTCOMES:
Minimal residual disease (MRD) | Up to 5 years
  MRD negative status and exploratory biomarkers will be summarized graphically and with descriptive statistics.
Association of biomarkers to overall response | Up to 5 years
  Association between molecular and cellular markers and overall response and/or resistance assessed through logistic regression analyses.
Change in markers over time | Baseline up to 5 years
  Paired t-test or Wilcoxon signed rank test will be used to assess the marker change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Venugopal S, Takahashi K, Daver N, Maiti A, Borthakur G, Loghavi S, Short NJ, Ohanian M, Masarova L, Issa G, Wang X, Carlos BR, Yilmaz M, Kadia T, Andreeff M, Ravandi F, Konopleva M, Kantarjian HM, DiNardo CD. Efficacy and safety of enasidenib and azacitidine combination in patients with IDH2 mutated acute myeloid leukemia and not eligible for intensive chemotherapy. Blood Cancer J. 2022 Jan 25;12(1):10. doi: 10.1038/s41408-021-00604-2. PMID 35078972
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org